CLINICAL TRIAL: NCT03120182
Title: Impact of Perioperative Maintenance or Interruption of Low-dose Aspirin on Recurrence Rate and Thrombotic Events After Burr-hole Drainage of Chronic Subdural Hematoma: a Randomized, Placebo Controlled, Double Blinded Study
Brief Title: Chronic Subdural Hematoma and Aspirin
Acronym: SECA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SECA
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Chronic Subdural Hematoma
Keywords: aspirin; bleeding risk; intracranial bleeding; burr-hole drainage; chronic subdural hematoma; anticoagulation
MeSH Terms: conditions — Hematoma, Subdural, Chronic; Intracranial Hemorrhages | interventions — Aspirin

STUDY DESIGN:
Intervention Model Description: randomized, placebo controlled, double blinded study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blinded study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aspirin Arm (Active Comparator): The patients will receive acetylsalicylic acid (100mg once a day, orally) for 12 days whereas the normal ASA treatment will be resumed 12 days after randomization
  Interventions: Drug: Acetylsalicylic acid
- Placebo Arm (Placebo Comparator): The patients will receive placebo oral tablets for 12 days whereas the normal ASA treatment will be resumed 12 days after randomization
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Acetylsalicylic acid — Patients will receive acetylsalicylic acid 100mg daily for 12 days after randomization
  Other Names: Aspirin
  Arms: Aspirin Arm
Drug: Placebo Oral Tablet — Patients will receive placebo medication 100mg daily for 12 days after randomization
  Other Names: Placebo
  Arms: Placebo Arm

SUMMARY:
The aim of this randomized, blinded, placebo controlled clinical study is to compare the peri- and postoperative bleeding and cardiovascular complication rates of patients undergoing burr-hole trepanation for chronic subdural hematoma with and without discontinuation of low-dose aspirin

DETAILED DESCRIPTION:
Chronic subdural hematoma (cSDH) is one of the most common neurosurgical conditions. Its significantly higher prevalence among patients older than 65 (69%) versus younger (31%) explains why 41% of the patients are taking blood thinners. Antiplatelet therapy in patients with chronic subdural hematoma (cSDH) presents significant neurosurgical challenges. Studies investigating the effect of acetylsalicylic acid (ASA) in cranial neurosurgery are sparse and mostly based on case reports. Given the lack of guidelines regarding perioperative management with antiplatelet therapy, it is difficult to balance the patient's increased cardiovascular risk and prevalence of cSDH. The aim of our randomized, blinded, placebo controlled clinical study is to compare the peri- and postoperative bleeding and cardiovascular complication rates of patients undergoing burr-hole trepanation for cSDH with and without discontinuation of low-dose ASA. We will include patients receiving low-dose ASA as secondary prophylaxis for various reasons (e.g. coronary artery disease (CAD), cerebrovascular disease, etc.) and will randomize them either to a Placebo- or Aspirin-arm. The patients will receive placebo or ASA for 12 days whereas the normal ASA treatment will be resumed 12 days after randomization. Our study primarily seeks to evaluate the risk of recurrence after burr-hole trepanation for cSDH under low-dose ASA treatment compared to placebo treatment. Secondary objectives are to assess the rate of thrombotic events, perioperative blood loss, postoperative anemia, intra- and postoperative blood transfusion rate, and clinical outcome (mRS, GOS, Markwalder score). The study will be performed in cooperation with the Department of Cardiology of the University Hospital of Basel.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing burr hole trepanation for cSDH who are under low-dose aspirin treatment ( Aspirin cardio 100mg once a day) for secondary prophylaxis

Exclusion Criteria:

* Patients under the age of 18years
* A recent (30 days before randomization) major cardiac event (i.e. unstable angina, myocardial infarction, or coronary revascularization)
* A recent (30 days before randomization) active bleeding event.
* Patient with known bleeding disorder (e.g. hemophilia)
* No informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2018-02-19 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Revision surgery due to a recurrent subdural hematoma | 6 months
  Recurrence of chronic subdural hematoma requiring revision surgery (burr-hole drainage)

SECONDARY OUTCOMES:
Myocardial infarction | 6 months
  (STEMI/non-STEMI)
Stroke | 6 months
  cerebral stroke
Peripheral arterial occlusion | 6 months
  occlusion of a peripheral artery
Other bleeding events apart from recurrent chronic subdural hematoma managed operatively or conservatively | 6 months
  acute subdural hematoma (aSDH), acute epidural hematoma (EDH), intraparenchymal bleeding)
Intraoperative blood loss | on the operation day (up to 1 day)
  blood loss recorded during surgery
Amount of blood/ fluid collected in the drain | up to 2 days, at removal of the drainage
  Amount of blood/ fluid collected in the drain
Postoperative anemia | up to 7 days
  hemoglobin<80mg/L
Operation time | during surgery
  Operation time
Hospitalization time | an average of 7 days
  Hospitalization time
Intraoperative blood transfusion rate | during surgery (e.g. up to 1 day)
  blood transfusion rate intraoperatively
Postoperative blood transfusion rate | during hospitalization, an average of 7 days
  blood transfusion rate postoperatively
GCS Score | 6 months
  Glasgow Coma Scale
mRS | 6 months
  modified Rankin scale
GOS | 6 months
  Glasgow Outcome Scale
Clinical outcome | 6 months
  Markwalder Score

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Mariani, Prof, MD, Study Chair — Department of Neurosurgery, University Hospital Basel; Maria Kamenova, MD, Principal Investigator — Department of Neurosurgery, University Hospital Basel; Jehuda Soleman, MD, Principal Investigator — Department of Neurosurgery, University Hospital Basel
Locations (1):
- Department of Neurosurgery, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kamenova M, Pacan L, Mueller C, Coslovsky M, Lutz K, Marbacher S, Moser M, Hickmann AK, Zweifel C, Guzman R, Mariani L, Soleman J; SECA Investigators. Aspirin Continuation or Discontinuation in Surgically Treated Chronic Subdural Hematoma: A Randomized Clinical Trial. JAMA Neurol. 2025 Jun 1;82(6):551-559. doi: 10.1001/jamaneurol.2025.0850. PMID 40287938
- [Derived] Kamenova M, Mueller C, Coslovsky M, Guzman R, Mariani L, Soleman J. Low-dose aspirin and burr-hole drainage of chronic subdural hematoma: study protocol for a randomized controlled study. Trials. 2019 Jan 21;20(1):70. doi: 10.1186/s13063-018-3064-y. PMID 30665464